CLINICAL TRIAL: NCT03710616
Title: A Real-world Study to Explore Recurrence/Metastases of the Early-stage (I-IIIA) NSCLC Patients and the Impact Factors of Patient Survivals
Brief Title: A Real-world Study to Explore Recurrence/Metastases of the NSCLC Patients and the Impact Factors of Patient Survivals
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Professor, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: GZH-001
Record Dates: First submitted 2018-07-10; First posted 2018-10-18 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Non-small Cell Lung Cancer
Keywords: early-stage NSCLC, real-world evidences, patient survivals
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Surgeries — Surgical operations plus systematic lymphadenectomies

SUMMARY:
The real-world study was designed to explore recurrence/metastases of the patients with non-small cell lung cancer as measured by patient survivals and the impact factors of patient survivals.

DETAILED DESCRIPTION:
The trial was designed as a real-world observational study to recruit those patients with pathologically diagnosed early-phase non-small cell lung cancer (NSCLC) who were enrolled in the clinical form 2009 to 2017 and explore recurrence/metastases of the NSCLC patients as measured by patient survivals and the impact factors of patient survivals. The study data on patient demographic characteristics, tumor biological characteristics, and clinicla treatments were collected via a retrospectively review method for evaluation of patient survivals and the relevance of clinical characteristics of the patients and patient survivals.

ELIGIBILITY:
Inclusion Criteria:

The patients who meet all the following inclusion criteria will be included in the study:

* The patients who were operated with radical operations of the lung cancer;
* The patients with clinical I-IIIA staging tumors;
* The pathologically diagnosed NSCLC patients;

Exclusion Criteria:

- Not be specified;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pathologically diagnosed early-stage (I-IIIA) NSCLC patients who were operated with radical operations of the lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2018-03-24 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival rates within the configured observation periods | 2009-2017
  Disease-free survival rates within 3-month, 6-month, 1-year, 2-year, and 3-year observation periods;

SECONDARY OUTCOMES:
Disease-free survival rates at the configured locations and observation periods | 2009-2017
  Disease-free survival rates at the metastasized lymph nodes, bone, and brain within 3-month, 6-month, 1-year, 2-year, and 3-year observation periods;

OTHER OUTCOMES:
Impact factors of disease-free survival rates | 2009-2017
  Impact factors of disease-free survival rates
Overall rates | 2009-2017
  Overall rates within 3 month-, 6 month-, 1 year-, 2 year-, and 3 year- observation periods
Rates of perioperative complications | 2009-2017
  Rates of perioperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Wenhua LIANG, Ph.D, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Department of Thoracic Surgery, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No